CLINICAL TRIAL: NCT01617837
Title: The Efficacy of P6 Acupressure in Reducing Postoperative Nausea and Vomiting in Patients Undergoing Craniotomy. - a Randomized, Double-blinded, Placebo Controlled Study.
Brief Title: The Efficacy of P6 Acupressure in Reducing Postoperative Nausea and Vomiting in Patients Undergoing Craniotomy
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Umeå University (Other)
Responsible Party: Principal Investigator, Ulrica G Nilsson, PhD, Associate Professor, Umeå University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2011-281-31M
Record Dates: First submitted 2012-06-09; First posted 2012-06-12 (Estimated); Last update posted 2013-09-18 (Estimated); Status verified 2013-09

CONDITIONS: Postoperative Nausea and Vomiting; Acupressure; Craniotomy
Keywords: Postoperative nausea and vomiting; P6 acupressure; Craniotomy.
MeSH Terms: conditions — Postoperative Nausea and Vomiting

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- P6 acupressure group (Active Comparator): In the end of the operation Sea-Band®, a single-sized elastic acupressure band with a plastic button, was placed unilaterally at the place of P6 (the P6 "Neiguan" acupoint, located about 3 cm proximal to the distal wrist, between the tendons of the flexor carpi radialis and the palmaris longus)to apply acupressure.
  Interventions: Device: P6 acupressure band
- Placebo group (Placebo Comparator): In the end of the operation an identical Sea-Band® with no button and thereby no acupressure was placed unilaterally at the place of P6.
  Interventions: Other: Placebo band

INTERVENTIONS:
Device: P6 acupressure band — Comparison between groups 0-48 hours postoperatively.
  Other Names: Sea-Band®
  Arms: P6 acupressure group
Other: Placebo band — Comparison between groups 0-48 hours postoperatively
  Other Names: Sea-Band® with no acupressure
  Arms: Placebo group

SUMMARY:
The aim of this study is to investigate if P6 acupressure may reduce postoperative nausea and vomiting in neurosurgical patients undergoing craniotomy.

DETAILED DESCRIPTION:
The primary aim of this study is to investigate if P6 acupressure can reduce postoperative nausea after craniotomy. Calculation of sample size was based on the assumptions to detect at difference of 20% between the patients (38% in the control group vs 18% in the acupressure group) for the primary endpoint; incidence of nausea during the first 24 hours postoperatively, with a significance level 5% and a power of 80%, guided by an earlier study with a similar population (Wang et. al. 2010) and the assumption that 38% of our patients suffer from nausea. These assumptions suggested a sample size of 78 patients (39 patients / group) that resulted in a sample size of 80 patients for covering attrition. Secondary aims are to investigate if the frequency of vomiting and the need for antiemetic can be reduced with P6 acupressure.

Patients are randomly assigned into one of two treatment groups using a computer-generated random number table, either P6 acupressure group or placebo group. Randomization and sealing of the study envelopes, containing all study material and following the patients all through the study, are performed by persons from the research department, who is not involved in the data collection. Information and study protocol are included in the envelope. The randomization is taking place preoperatively. Sea-Band®, a single-sized elastic acupressure band with a plastic button placed at P6 to apply pressure is used. One group will receive an active acupressure band and the other an identical placebo band without any button. Before entering the operation ward both wrists are marked at the place for P6, performed by staff at the neurosurgical ward. The active acupressure bands and the placebo bands are administered at the end of surgery. They are placed unilaterally at the wrist by the nurse anesthetist who performs the patient's anesthesia. The manufacturer's guidelines of where and how to place the band are included in the envelope with study material. Both the P6 acupressure bands and the placebo bands are covered with a bandage to ensure blinding to the patients and the nursing staff involved in the postoperative care. Both the P6 acupressure bands and the placebo bands will be removed 48 hours postoperatively. If the bands cause discomfort, they can be removed for 30 minutes every two hours, performed by staff not involved in the postoperative care, with instructions to cover the wrist with a cotton roll while airing the arm, this for ensuring further blinding if the acupressure has caused any betrayal marks.

At the end of the surgery all patients receive ondansetron 4mg IV. Droperidol IV is administered as additional perioperative antiemetic if considered necessary. Postoperatively rescue antiemetics are administrated according to current routines. The administered drugs are 0,625-1,25mg droperidol and 1-4mg ondansetron, either alone or in combination. Postoperative opioid administration (morphine and ketobemidone) are also recorded during the time of the study

Before operation all patients are filling in a health declare formula as a routine in the anesthetic preparation. This formula includes the four risk factors for PONV, according to Apfel and colleagues (Apfel et al. 1999). To clarify earlier PONV there is a specific question about this issue on the formula of written consent.

During 48 hours postoperatively the patients are evaluating their nausea which is registered on the same formula as the frequencies of vomiting. The first evaluation is taking part when arriving to the postoperative care unit and then every hour for the first six hours, every third hour until hour 24 and thereafter every sixth hour from hour 25-48. A Numerical Rating Scale (NRS) from 0-10 is used, where 0 mean no nausea at all and 10 the worst nausea possible. The patients are asked about whether they have experienced any nausea within the previous period of time. Assessment of nausea and registration of the vomiting frequency are performed by staff unaware of the patient's group in the postoperative care unit/neurosurgical ward and by the patients themselves when possible.

After discharge the data from the NRS formula are collected. The patients' journals are screened for administrated antiemetic and opioids, for potential risk factors for PONV and for other demographics relevant to the study outcome. All data are saved anonymously in the software Statistical Package for Social Sciences (SPSS).

Overall PONV is defined as at least one episode of nausea or vomiting during the observation time of 48 h. Rescue therapy is defined as at least one dosage of either droperidol or ondansetron during the observation time of 48 h. Early PONV is defined as PONV occurring up to 6 hours postoperatively and late PONV 7-48 hours postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* Elective infra-or supratentorial craniotomy
* Age ≥ 18 years

Exclusion Criteria:

* Patients not able to actively participate in the study according to mental status or communicating problems and patients receiving an antiemetic less than twelve hours before surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2011-11; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Postoperative nausea and vomiting | Postperative nauea and vomiting are registred regularly 0-48 hours postperatively.
  During 48 hours postoperatively the patients are evaluating their nausea, registered on the same formula as the frequencies of vomiting. The first evaluation will take part when arriving to the postoperative care unit and then every hour for the first six hours, every third hour until hour 24 and thereafter every sixth hour from hour 24-48. A Numerical Rating Scale (NRS) from 0-10 will be used, where 0 means no nausea at all and 10 the worst nausea possible. The patients will be asked about whether they have experienced any nausea within the previous period of time.

CONTACTS AND LOCATIONS:
Overall Officials: Ulrica Nilsson, PhD, Study Director — Umeå University
Locations (1):
- The Department of Neurosurgery, Umeå University Hospital, Umeå, Västerbotten County, Sweden